CLINICAL TRIAL: NCT06934109
Title: Acceptability and Feasibility of an Adapted Narrative Exposure Therapy (NET) Protocol for Individuals With an Intellectual Disability
Brief Title: Narrative Exposure Therapy for Adults With an Intellectual Disability
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24042
Record Dates: First submitted 2025-02-26; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Trauma, Psychological; Learning Disability; PTSD; Intellectual Disability, Mild
MeSH Terms: conditions — Psychological Trauma; Learning Disabilities; Stress Disorders, Post-Traumatic; Intellectual Disability; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Narrative Exposure Therapy treatment (Experimental): All participants within the trial will receive narrative exposure therapy and be within the treatment arm.
  Interventions: Other: Narrative Exposure Therapy (NET)

INTERVENTIONS:
Other: Narrative Exposure Therapy (NET) — NET is a psychological talking therapy that has been designed for people who have experienced multiple and prolonged traumatic experiences. It is typically 12-sessions, involving first a psychoeducation session, then laying a lifeline where stones are lain to represent traumatic events, and flowers positive life events. The following sessions the person is asked to talk through their life, going into detail on the traumatic memories that they have experienced.

SUMMARY:
The goal of this naturalistic single case series design is to investigate if an adapted Narrative Exposure Therapy protocol can be effective, is feasible, and acceptable for adults with a mile learning disability.

Participants will be complete three baseline sessions before taking part in Narrative Exposure Therapy using a manual that has been adapted for people with a learning disability. Trauma symptoms will be measured weekly using the Impact of Events scale adapted for intellectual disabilities. The person's carer will also complete an informant scale related to these symptoms (LANTS-IV). The client will also complete the CORE-LD at pre, and post therapy. Six weeks after the end of the intervention, the client and their carer will be invited to a feedback session to talk about how they found the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Meet the criteria for having a mild ID as assessed by a clinical psychologist within the team
* English speaking
* Have capacity to consent
* The participant must be experiencing trauma related stress as assessed by themselves, the clinical psychologist and the research team
* Be able to travel to one of the therapy sites
* Carer participant must have ability to reflect and comment on the trauma related stress experienced by the client participant
* Carer must also be 18 years old or older and be English speaking.
* Carer must have known participant for 1 year or more.

Exclusion Criteria:

* They are substance dependent
* They are currently receiving another trauma-focused intervention
* Currently an inpatient
* Carers excluded if they lack capacity to consent to take part in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Impact of Events Scale for intellectual disabilities (IES-ID) | Completed weekly through baseline and intervention stages, approximately 16 weeks. Then at 6-week follow up (approximately week 22).
  The IES-ID (Hall et al., 2014) is a 22 item scale scored on a three-point Likert scale measuring trauma related symptoms. This is an adapted measure that has been validated for people with an intellectual disability.
Lancaster and Northgate Trauma Scale for Intellectual Disabilities - Informant Version (LANTS-IV; Wigham et al., 2011) | Completed weekly through baseline and intervention stages, approximately 16 weeks. Then at 6-week follow up (approximately week 22).
  47 scored on a six-point scale for frequency and three-point for severity.
Clinical Outcome Routine Evaluation-Learning Disabilities (CORE-LD; Brooks et al., 2013) | At baseline week 1 and at 6-week follow-up (approximately week 22).
  14 scored on a three-point Likert scale measuring psychological distress across four domains: well-being, symptoms, functioning, and risk
Change interview (Elliott et al., 2001) with clients and carers | 6-weeks post-intervention. Sessions will be around 30-60 minutes.
  A feedback session will be held with the client and their carer around 6-weeks after the therapy has come to an end. This will ask for feedback on how they found the intervention.

SECONDARY OUTCOMES:
Heart rate | Weekly during the intervention sessions, for approximately 12-weeks.
  Heart rate will be taken using a fitness watch that can measure continuous heart rate. This will show whether any within and between session habituation has taken place. Subjective units of distress (Wolpe, 1969) will be used if clients do not wish to wear a heart rate device.
Post-session therapist reflections | Across the intervention phase, an average of a year
  Therapist reflections will be collected to gather information about their thoughts relating to the manual and therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schroder, Principal Investigator — University of Nottingham
Locations (1):
- Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, United Kingdom